CLINICAL TRIAL: NCT02820324
Title: A Phase 3, Multicenter, Randomized, Double-Blind, Placebo and Active-Controlled Study of Oliceridine (TRV130) for the Treatment of Moderate to Severe Acute Pain After Abdominoplasty
Brief Title: Study of Oliceridine (TRV130) for the Treatment of Moderate to Severe Acute Pain After Abdominoplasty
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Trevena Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CP130-3002
Record Dates: First submitted 2016-06-09; First posted 2016-06-30 (Estimated); Results first posted 2020-10-23 (Actual); Last update posted 2020-10-23 (Actual); Status verified 2020-09

CONDITIONS: Acute Pain
MeSH Terms: conditions — Acute Pain | interventions — ((3-methoxythiophen-2-yl)methyl)((2-(9-(pyridin-2-yl)-6-oxaspiro(4.5)decan-9-yl)ethyl))amine; Morphine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (5):
- Treatment 1 Oliceridine (Experimental)
  Interventions: Drug: Oliceridine
- Treatment 2 Oliceridine (Experimental)
  Interventions: Drug: Oliceridine
- Treatment 3 Oliceridine (Experimental)
  Interventions: Drug: Oliceridine
- Treatment 4 Placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- Treatment 5 Morphine (Active Comparator)
  Interventions: Drug: Morphine

INTERVENTIONS:
Drug: Oliceridine
  Arms: Treatment 1 Oliceridine; Treatment 2 Oliceridine; Treatment 3 Oliceridine
Drug: Placebo
  Arms: Treatment 4 Placebo
Drug: Morphine
  Arms: Treatment 5 Morphine

SUMMARY:
The primary objective is to evaluate the analgesic efficacy of intravenous (IV) oliceridine administered as needed (PRN) compared with placebo in patients with moderate to severe acute pain after abdominoplasty.

ELIGIBILITY:
Inclusion Criteria:

* Has undergone abdominoplasty with no additional collateral procedures.
* Experiences a pain intensity rating of moderate to severe acute pain.
* Able to provide written informed consent before any study procedure.

Exclusion Criteria:

* ASA Physical Status Classification System classification of P3 or worse.
* Has surgical or post-surgical complications.
* Has clinically significant medical conditions or history of such conditions that may interfere with the interpretation of efficacy, safety, or tolerability data obtained in the trial, or may interfere with the absorption, distribution, metabolism, or excretion of drugs.
* Has previously participated in another TRV130 clinical study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 407 (Actual)
Dates: Start 2016-05; Primary Completion 2016-12 (Actual); Study Completion 2017-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Franck Skobieranda, MD, Study Director — Trevena Inc.
Locations (5):
- United States (5):
  - Research Site, Phoenix, Arizona
  - Research Site, Pasadena, California
  - Research Site, Pasadena, Maryland
  - Research Site, Houston, Texas
  - Research Site, San Antonio, Texas

REFERENCES:
- [Derived] Singla NK, Skobieranda F, Soergel DG, Salamea M, Burt DA, Demitrack MA, Viscusi ER. APOLLO-2: A Randomized, Placebo and Active-Controlled Phase III Study Investigating Oliceridine (TRV130), a G Protein-Biased Ligand at the mu-Opioid Receptor, for Management of Moderate to Severe Acute Pain Following Abdominoplasty. Pain Pract. 2019 Sep;19(7):715-731. doi: 10.1111/papr.12801. Epub 2019 Jun 24. PMID 31162798

RESULTS

PARTICIPANT FLOW:
Groups:
- Treatment 1 Oliceridine: Oliceridine 0.1 mg
  The loading dose was 1.5 mg with PCA demand doses of 0.1 mg. Supplemental doses of 0.75 mg were permitted, beginning 1 hour after the loading dose, and hourly thereafter, as needed. A lockout interval of 6 minutes was used for all PCA regimens.
- Treatment 2 Oliceridine: Oliceridine 0.35 mg
  The loading dose was 1.5 mg with PCA demand doses of 0.35 mg. Supplemental doses of 0.75 mg were permitted, beginning 1 hour after the loading dose, and hourly thereafter, as needed. A lockout interval of 6 minutes was used for all PCA regimens.
- Treatment 3 Oliceridine: Oliceridine 0.5 mg
  The loading dose was 1.5 mg with PCA demand doses of 0.5 mg. Supplemental doses of 0.75 mg were permitted, beginning 1 hour after the loading dose, and hourly thereafter, as needed. A lockout interval of 6 minutes was used for all PCA regimens.
- Treatment 4 Placebo: Placebo
  The loading dose was 1.5 mL with volume-matched PCA demand doses. Supplemental doses of 0.75 mL were permitted, beginning 1 hour after the loading dose, and hourly thereafter, as needed. A lockout interval of 6 minutes was used for all PCA regimens.
- Treatment 5 Morphine: Morphine
  The loading dose for the morphine treatment regimen was 4 mg with 1 mg demand doses. Supplemental doses of 2 mg were permitted, beginning 1 hour after the loading dose, and hourly thereafter, as needed. A lockout interval of 6 minutes was used for all PCA regimens.
Period: Overall Study
Arm/Group | Treatment 1 Oliceridine | Treatment 2 Oliceridine | Treatment 3 Oliceridine | Treatment 4 Placebo | Treatment 5 Morphine
Started | 78 | 82 | 82 | 82 | 83
Treated With Study Medication | 77 | 80 | 80 | 81 | 83
Completed | 76 | 79 | 79 | 79 | 80
Not Completed | 2 | 3 | 3 | 3 | 3

BASELINE CHARACTERISTICS:
Groups:
- Treatment 1 Oliceridine: Oliceridine 0.1 mg
- Treatment 2 Oliceridine: Oliceridine 0.35 mg
- Treatment 3 Oliceridine: Oliceridine 0.5 mg
- Treatment 4 Placebo: Placebo
- Treatment 5 Morphine: Morphine
- Total: Total of all reporting groups
Arm/Group | Treatment 1 Oliceridine | Treatment 2 Oliceridine | Treatment 3 Oliceridine | Treatment 4 Placebo | Treatment 5 Morphine | Total
Number analyzed (Participants) | 77 | 80 | 80 | 81 | 83 | 401
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 74 | 78 | 79 | 79 | 81 | 391
  >=65 years | 3 | 2 | 1 | 2 | 2 | 10
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.8 (10.64) | 42 (9.97) | 40.4 (10.03) | 42.2 (10.25) | 40.4 (10.35) | 41.4 (10.23)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 76 | 80 | 80 | 81 | 81 | 398
  Male | 1 | 0 | 0 | 0 | 2 | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 28 | 24 | 24 | 27 | 29 | 132
  Not Hispanic or Latino | 49 | 56 | 56 | 54 | 54 | 269
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 0 | 0 | 0 | 1
  Asian | 3 | 2 | 1 | 1 | 2 | 9
  Native Hawaiian or Other Pacific Islander | 2 | 0 | 0 | 0 | 1 | 3
  Black or African American | 24 | 22 | 28 | 27 | 24 | 125
  White | 45 | 55 | 50 | 52 | 55 | 257
  More than one race | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 2 | 1 | 1 | 1 | 1 | 6
Region of Enrollment [Number; unit: participants]
  United States | 77 | 80 | 80 | 81 | 83 | 401

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients Who Respond to Study Medication at the 24-hr Numeric Pain Rating Scale (NPRS) Assessment Compared to Placebo.
Description: The NPRS is an 11-point scale from 0-10 where "0" = no pain and "10" = the most intense pain imaginable. A patient was a responder if: their final time-weighted Sum of Pain Intensity Difference (SPID)-24 corresponded to a ≥30% improvement without rescue pain medication during the Randomized Treatment Period, without early discontinuation of study medication for any reason, and without reaching the study medication dosing limit.
Time Frame: 24 hours
Population: The analysis population reflects the number of patients treated with study medication.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment 1 Oliceridine | Treatment 2 Oliceridine | Treatment 3 Oliceridine | Treatment 4 Placebo | Treatment 5 Morphine
Number analyzed (Participants) | 77 | 80 | 80 | 81 | 83
Participants | 47 | 61 | 56 | 37 | 65

2. Secondary Outcome: Number of Respiratory Safety Events Compared to Morphine.
Description: Respiratory Safety Events were defined as a clinically relevant worsening of respiratory status.
Time Frame: 24 hours
Population: The analysis population reflects the number of patients treated with study medication.
Measure: Number; unit: Respiratory Safety Events
Arm/Group | Treatment 1 Oliceridine | Treatment 2 Oliceridine | Treatment 3 Oliceridine | Treatment 4 Placebo | Treatment 5 Morphine
Number analyzed (Participants) | 77 | 80 | 80 | 81 | 83
Respiratory Safety Events | 6 | 17 | 18 | 5 | 22

3. Secondary Outcome: Duration of Respiratory Events Compared to Morphine.
Description: Respiratory Safety Events were defined as a clinically relevant worsening of respiratory status.
Time Frame: 24 hours
Population: The analysis population reflects the number of patients treated with study medication.
Measure: Mean (Standard Error); unit: hours
Arm/Group | Treatment 1 Oliceridine | Treatment 2 Oliceridine | Treatment 3 Oliceridine | Treatment 4 Placebo | Treatment 5 Morphine
Number analyzed (Participants) | 77 | 80 | 80 | 81 | 83
hours | 2.27 (0.924) | 2.97 (0.815) | 3.43 (1.049) | 4.12 (1.687) | 3.17 (0.869)

4. Secondary Outcome: Odds Ratio of Patients Who Respond to Study Medication at the 24-hr NPRS Assessment Compared to Morphine.
Description: Odds ratio of 24-hour responder analysis versus morphine. Number of patients who responded to study medication at the 24-hr NPRS assessment is captured in the primary outcome measure.
Time Frame: 24 hours
Population: The analysis population reflects the number of patients treated with study medication. The morphine and placebo Arms/Groups are not included, as this is a comparison of study medication against morphine.
Measure: Number; unit: odds ratio
Arm/Group | Treatment 1 Oliceridine | Treatment 2 Oliceridine | Treatment 3 Oliceridine
Number analyzed (Participants) | 77 | 80 | 80
odds ratio | 0.88 | 2.11 | 1.73

5. Secondary Outcome: Number of Patients With Treatment-related Adverse Events Compared to Placebo and Compared to Morphine.
Time Frame: 24 hours
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment 1 Oliceridine | Treatment 2 Oliceridine | Treatment 3 Oliceridine | Treatment 4 Placebo | Treatment 5 Morphine
Number analyzed (Participants) | 77 | 80 | 80 | 81 | 83
Participants | 52 | 70 | 70 | 44 | 76

ADVERSE EVENTS:
Arm/Group | Treatment 1 Oliceridine | Treatment 2 Oliceridine | Treatment 3 Oliceridine | Treatment 4 Placebo | Treatment 5 Morphine
All-Cause Mortality (participants affected / at risk) | 0/77 | 0/80 | 0/80 | 0/81 | 0/83
Serious Adverse Events (participants affected / at risk) | 0/77 | 1/80 | 3/80 | 0/81 | 1/83
Other Adverse Events (participants affected / at risk) | 69/77 | 74/80 | 76/80 | 65/81 | 80/83
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment 1 Oliceridine (N=77) | Treatment 2 Oliceridine (N=80) | Treatment 3 Oliceridine (N=80) | Treatment 4 Placebo (N=81) | Treatment 5 Morphine (N=83)
Abdominal Wall Hematoma (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Post Procedural Hemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lethargy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment 1 Oliceridine (N=77) | Treatment 2 Oliceridine (N=80) | Treatment 3 Oliceridine (N=80) | Treatment 4 Placebo (N=81) | Treatment 5 Morphine (N=83)
Nausea (Gastrointestinal disorders) | 34 | 49 | 60 | 38 | 61
Vomiting (Gastrointestinal disorders) | 18 | 17 | 34 | 11 | 44
Headache (Nervous system disorders) | 12 | 23 | 21 | 24 | 24
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 6 | 16 | 14 | 4 | 19
Constipation (Gastrointestinal disorders) | 12 | 13 | 9 | 6 | 9
Pruritus (Skin and subcutaneous tissue disorders) | 10 | 13 | 9 | 4 | 15
Dizziness (Nervous system disorders) | 11 | 7 | 7 | 9 | 13
Sedation (Nervous system disorders) | 5 | 11 | 7 | 7 | 19
Back Pain (Musculoskeletal and connective tissue disorders) | 3 | 10 | 9 | 5 | 7
Hot Flash (Vascular disorders) | 2 | 6 | 5 | 6 | 6
Anxiety (Psychiatric disorders) | 1 | 4 | 6 | 2 | 3
Rash (Skin and subcutaneous tissue disorders) | 3 | 1 | 6 | 2 | 0
Restlessness (Psychiatric disorders) | 1 | 5 | 3 | 3 | 4
Hyperhydrosis (Skin and subcutaneous tissue disorders) | 2 | 4 | 2 | 2 | 2
Pruritus Generalized (Skin and subcutaneous tissue disorders) | 1 | 1 | 6 | 1 | 7
Myalgia (Musculoskeletal and connective tissue disorders) | 2 | 4 | 1 | 1 | 0
Abdominal Pain Upper (Gastrointestinal disorders) | 5 | 1 | 0 | 3 | 2
Flatulence (Gastrointestinal disorders) | 4 | 1 | 1 | 4 | 2
Presyncope (Nervous system disorders) | 4 | 1 | 1 | 0 | 2
Somnolence (Nervous system disorders) | 2 | 0 | 4 | 1 | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other